CLINICAL TRIAL: NCT06864039
Title: Quality of Life and Long-term Outcome of Transition-age Patients With Congenital Hypothyroidism Diagnosed by Newborn Screening and Adequately Treated
Brief Title: Quality of Life and Long-term Outcome of Adequately Treated Congenital Hypothyroidism
Acronym: CHQoL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof.ssa Mariacarolina Salerno, Full Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 245/2023
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Congenital Hypothyroidism
Keywords: quality of life; congenital hypothyroidism; treatment; newborn screening; outcome
MeSH Terms: conditions — Congenital Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adolescents aged 16-21 years with congenital hypothyroidism diagnosed by newborn screening (Other): A) Clinical assessment (Weight, Height, BMI, Waist and hip circumference, blood pressure) B) Assessment of body composition by performing bioimpedance analysis C) Assessment of quality of life by administering the SF36 test D) Assessment of cognitive abilities by administering the WAIS IV test E) Assessment of any psychopathological conditions by means of the SCL-90 psychopathological screening questionnaire F) For patients up to 18 years of age: CBCL questionnaire to be administered to parents to assess the patient's behavior
  Interventions: Diagnostic Test: SF36 test; Diagnostic Test: WAIS IV test; Diagnostic Test: SCL-90 psychopathological screening questionnaire; Diagnostic Test: CBCL questionnaire; Diagnostic Test: bioimpedance analysis

INTERVENTIONS:
Diagnostic Test: SF36 test — Assessment of quality of life by administering the SF36 test
Diagnostic Test: WAIS IV test — Assessment of cognitive abilities by administering the WAIS IV test
Diagnostic Test: SCL-90 psychopathological screening questionnaire — Assessment of any psychopathological conditions by means of the SCL-90 psychopathological screening questionnaire
Diagnostic Test: CBCL questionnaire — For patients up to 18 years of age: CBCL questionnaire to be administered to parents to describe the patient's behavior
Diagnostic Test: bioimpedance analysis — Assessment of body composition by performing bioimpedance analysis

SUMMARY:
The primary objective of this observational study is the evaluation of the quality of life and long-term outccome of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening receiving replacement treatment with levothyroxine.

The secondary objective is to relate the results to the form of hypothyroidism, the initial dose of L-T4, treatment adherence and genetics

DETAILED DESCRIPTION:
The study protocol will be performed in 3 different phases:

Step1:

A) Enrollment of patients meeting the following criteria:

* diagnosis of congenital hypothyroidism through neonatal screening adequately treated with L-T4
* confirmation of the diagnosis of hypothyroidism upon re-evaluation of the diagnosis
* age 16-21 years at the time of enrollment

B) Information interview on the study and signing of informed consent by the patient and/or parent/guardian

C) Retrospective collection of the following parameters at diagnosis:

* Values of TSH, FT4 at diagnosis, initial dose of L-T4
* Thyroid ultrasound and scintigraphy reports
* Genetic investigation report if available

D) Retrospective collection for each year of follow-up of:

weight, height, TSH, FT4 and L-T4 dose

Step 2:

A) Clinical evaluation (Weight, Height, BMI, Waist and hip circumference, blood pressure) B) Evaluation of body composition by performing bioimpedance analysis C) Evaluation of quality of life through administration of the SF36 test D) Evaluation of cognitive abilities through administration of the WAIS IV test E) Evaluation of any psychopathological conditions through the SCL-90 psychopathological screening questionnaire F) For patients up to 18 years of age: CBCL questionnaire administered to parents to describe the patient's behaviour

Step 3:

Data collection and analysis of results

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital hypothyroidism by neonatal screening
* Start of L-T4 therapy within the first month of life
* Confirmation of hypothyroidism condition upon reassessment of diagnosis

Exclusion Criteria:

* other chronic diseases and/or genetic syndromes
* family history of neuropsychiatric pathology
* familial dyslipidemia

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening on levothyroxine replacement treatment. | evaluation of the long term outcomes at the time of enrolment
  Administration of the SF36 questionnaire for the evaluation of quality of life in transition-age children with adequately treated congenital hypothyroidism
Auxological outcome of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening on levothyroxine replacement treatment. | evaluation of the long term outcomes at the time of enrolment
  weigh SDS, height SDS and BMI SDS assessment in transition-age children with adequately treated congenital hypothyroidism
Intellectual outcome of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening on levothyroxine replacement treatment. | evaluation of the long term outcomes at the time of enrolment
  Assessment of cognitive abilities through the administration of the WAIS IV
Psychopathological condition of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening on levothyroxine replacement treatment. | evaluation of the long term outcomes at the time of enrolment
  Assessment of psychopathological conditions through the SCL-90 questionnaire
Behovioral outcome of young-adult patients with congenital hypothyroidism diagnosed by neonatal screening on levothyroxine replacement treatment. | evaluation of the long term outcomes at the time of enrolment
  Administration of the CBCL questionnaire to parents of patients up to 18 years of age to describe the patient's behavior

SECONDARY OUTCOMES:
Correlation between quality of life and type of congenital hypothyroidism | at time of enrollment
  Correlation between quality of life and type of congenital hypothyroidism with Pearson's test
Correlation between intellectual outcome and type of congenital hypothyroidism | at time of enrollment
  Correlation between intellectual outcome and type of congenital hypothyroidism with Pearson's test
Correlation between psychopathological evaluation and type of congenital hypothyroidism | at time of enrollment
  Correlation between psychopathological evaluation and type of congenital hypothyroidism with Pearson's test
Correlation between behovioral evaluation and type of congenital hypothyroidism | at time of enrollment
  Correlation between behovioral evaluation and type of congenital hypothyroidism with Pearson's test

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Endocrinology Program, Department of the Mother and the Child, University Federico II of Naples, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leger J, Ecosse E, Roussey M, Lanoe JL, Larroque B; French Congenital Hypothyroidism Study Group. Subtle health impairment and socioeducational attainment in young adult patients with congenital hypothyroidism diagnosed by neonatal screening: a longitudinal population-based cohort study. J Clin Endocrinol Metab. 2011 Jun;96(6):1771-82. doi: 10.1210/jc.2010-2315. Epub 2011 Mar 9. PMID 21389139